CLINICAL TRIAL: NCT06472128
Title: Multi-Site Randomized Controlled Trial of a Novel Digital Application (DREAMLAND) to Improve Outcomes for Patients With Acute Myeloid Leukemia
Brief Title: Novel Digital Application for Patients With Acute Leukemia
Acronym: NAVIGATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-025; R01CA288550 (NIH)
Record Dates: First submitted 2024-06-09; First posted 2024-06-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Relapsed Adult Acute Myeloid Leukemia; Primary Refractory Acute Myeloid Leukemia; High Risk Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DREAMLAND (Experimental): DREAMLAND is a self-administered, multicomponent mobile psychological intervention application for patients to be used during their hospitalization for intensive chemotherapy.
  Interventions: Behavioral: DREAMLAND
- VITAL WELLNESS (Active Comparator): VITAL WELLNESS is a self-administered, multicomponent mobile application containing information on a range of physical health topics that guide patients through education about general wellness, nutrition, exercise, and cancer prevention.
  Interventions: Behavioral: VITAL WELLNESS

INTERVENTIONS:
Behavioral: DREAMLAND — Participants assigned to DREAMLAND will start using DREAMLAND during the first week of their hospitalization, with a suggested timeline of reviewing one module each week to complete the required modules by week 4 of their hospital stay.
  Arms: DREAMLAND
Behavioral: VITAL WELLNESS — Participants assigned to VITAL WELLNESS will start using VITAL WELLNESS during the first week of their hospitalization, with a suggested timeline of reviewing one module each week to complete the required modules by week 4 of their hospital stay.
  Arms: VITAL WELLNESS

SUMMARY:
This research study is evaluating to examine the efficacy of a novel a self-administered digital application (DREAMLAND) for improving patients' long-term quality of life and psychological outcomes for patients with acute myeloid leukemia undergoing intensive chemotherapy.

DETAILED DESCRIPTION:
Patients newly diagnosed with acute myeloid leukemia (AML) confront a sudden and life-threatening diagnosis, requiring an immediate disruption of their life and an urgent 4-6-week hospitalization to initiate intensive chemotherapy. During this hospitalization, they endure substantial physical symptoms due to the side-effects of chemotherapy, which negatively impact their quality of life. Importantly, patients also experience immense psychological distress as they struggle with the abrupt onset of illness, uncertainty regarding their prognosis, physical and social isolation during hospitalization, and complete loss of independence.

Despite the well-described psychological sequalae patients with AML experience, interventions to support them during this challenging hospitalization are limited. Moreover, limited availability of palliative care and mental health clinicians further hinders the scalability and dissemination of supportive care interventions to address the needs of all patients with AML. The investigators developed a self-administered novel digital app (DREAMLAND) for patients with AML undergoing intensive chemotherapy. DREAMLAND includes four modules that focus on: 1) supportive psychotherapy to help patients adjust to the shock of diagnosis; 2) psychoeducation to manage illness expectations; 3) psychosocial skill-building to promote effective coping; and 4) self-care. The investigators recently completed a pilot randomized trial demonstrating the feasibility of DREAMLAND and its promising efficacy for improving patient reported quality of life, anxiety, and depression symptoms, as well as self-efficacy and symptom burden, compared to usual care. Based on these findings, DREAMLAND received an FDA Breakthrough Device Designation as a promising digital therapeutic for AML.

The purpose of this study is to conduct a multi-site randomized trial of DREAMLAND versus VITAL WELLNESS (a physical health promotion control app) in 200 patients with AML undergoing intensive chemotherapy to: a) demonstrate the efficacy of DREAMLAND versus VITAL WELLNESS for improving patient-reported quality of life, and psychological distress; b) assess the impact of DREAMLAND on patient-reported symptom burden, coping, and self-efficacy; c) explore mediators and moderators of the intervention effect on patient-reported quality of life; and d) establish the generalizability of DREAMLAND across care settings.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients (age > 18 years) with a diagnosis of AML.
* Initiating treatment with either a) intensive chemotherapy (7+3) or modification of this regimen on a clinical trial, or a similar intensive regimen or b) hypomethylating agents (HMA) +/- additional agents or modification of this regimen on a clinical trial.
* Ability to comprehend and speak English as the digital apps are only available in English

Note: Patients newly diagnosed as well as those with relapsed/refractory AML initiating treatment with intensive or HMA-based chemotherapy will be eligible to participate.

Exclusion Criteria:

* Patients with a diagnosis of acute promyelocytic leukemia
* Patients with acute or unstable psychiatric or cognitive conditions which the treating clinicians believes prohibits informed consent or compliance with study procedures.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient reported quality of life (QOL) at day 20 as measured by the Functional Assessment of Cancer Therapy-Leukemia scale | Day +20
  To compare QOL at day +20 between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leukemia) at day 20.
  Higher scores on FACT-Leukemia (range 0-176) indicate a better QOL.

SECONDARY OUTCOMES:
Longitudinal patient reported quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-Leukemia scale | Up to 180 days
  To compare QOL longitudinally between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leukemia).
  Higher scores on FACT-Leukemia (range 0-176) indicate a better QOL.
Participant anxiety symptoms assessed by the Hospital Anxiety and Depression Scale | Up to 180 days
  To compare anxiety symptoms (both at day +20 and longitudinally) between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Hospital Anxiety and Depression Scale (HADS) anxiety subscale.
  Lower scores on HADS anxiety subscale indicate less anxiety (score: 0-7-Normal, 8-10-Mild, 11-15-Moderate, 16-21-Severe).
Participant depression symptoms as measured by the Hospital Anxiety Depression scale | Up to 180 days
  To compare depression symptoms both at day +20 and longitudinally between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Hospital Anxiety and Depression Scale (HADS).
  Lower scores on HADS depression subscale indicate absence of depression (score: 0-7-Normal, 8-10-Mild, 11-15-Moderate, 16-21-Severe).
Participant depressive syndrome as measured by the patient Health Qiestionnaire-9 scale | Up to 180 days
  To compare depressive syndrome symptoms both at day +20 and longitudinally between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Patient Health Questionnaire-9 (PHQ-9).
  Lower PHQ-9 scores indicate absence or minimal depression (score: 0-4 -None-minimal, 5-9-Mild, 10-14-Moderate, 15-19-Moderately Severe, 20-27-Severe).
Participant symptom burden a assessed by the Edmonton Symptom Assessment scale | Day +20
  To compare symptom burden at day +20 between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Edmonton Symptom Assessment Scale (ESAS-R).
  A higher ESAS-R score (total ranges from 0 to 60) indicates a higher physical symptom burden.
Participant post-traumatic stress symptoms as assessed by the Post-traumatic Stress Disorder Checklist Civilian Version. | Up to 180 days
  To compare post-traumatic stress symptoms (both at day +20 and longitudinally) between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Post-traumatic Stress Disorder Checklist-Civilian Version.
  Scores above 44 indicates possible PTSD (scores range from 17 to 85).

OTHER OUTCOMES:
Participant perceived ability to used adaptive coping as measured by the Measure of Current Status Part A | Up to 180 days
  To compare coping (both at day +20 and longitudinally) between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Measure of Current Status Part A (MOCS-A).
  Higher MOCS-A scores indicate higher perceived ability to use adaptive coping techniques (scores range from 0-52).
Participant self-efficacy level as measured by the Cancer Self-Efficacy scale | Up to 180 days
  To compare self-efficacy (both at day +20 and longitudinally) between those receiving DREAMLAND versus VITAL WELLNESS as measured by the Cancer Self-Efficacy scale (CASE).
  Higher CASE scores indicate higher levels of self-efficacy (scores range from 12 to 48).
Participant experience of application's usability as measured by the Systems Usability Scale | Day +60
  To explore participants´ usability of the apps at day +60 as measured by the System Usability Scale (SUS).
  Higher SUS scores indicate higher levels of usability (scored on a 0-100 scale).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center (FHCRC), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation